CLINICAL TRIAL: NCT03701659
Title: A Prospective, Multi-center Clinical Study of Palliative Transurethral Plasma Kinetic Resection of Prostate (TUPKRP) Combined With Endocrine Therapy for Advanced Prostate Cancer Complicated With Severe Lower Urinary Tract Symptoms
Brief Title: TUPKRP Combined With MAB Therapy for LUTS/PCa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xy3yyUrology01
Record Dates: First submitted 2018-10-03; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Advanced Prostate Cancer; Lower Urinary Tract Symptoms; Quality of Life; Overall Survival; Progression of Prostate Cancer
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TUPKRP+MAB Group (Experimental): These patient will be treated by TUPKRP and MAB.
  Interventions: Procedure: Surgery combinate with Endocrine therapy
- MAB Group (Active Comparator): These patient will be treated by MAB only.
  Interventions: Drug: Endocrine therapy

INTERVENTIONS:
Procedure: Surgery combinate with Endocrine therapy — TUPKRP is abbreviation of transurethral plasma kinetic resection of prostate, which is an effective treatment of bladder outlet obstruction for benign prostate hyperplasia. MAB is abbreviation of Maximal androgen blockade, which is a kind of endocrinotherapy for advanced prostate cancer.
  Arms: TUPKRP+MAB Group
Drug: Endocrine therapy — MAB is abbreviation of Maximal androgen blockade, which is a kind of endocrine therapy for advanced prostate cancer.
  Arms: MAB Group

SUMMARY:
Prostate cancer (PCa) is the second most frequently diagnosed cancer in men worldwide, accounting for 15% of all male cancers. In 2015, there were 220,800 estimated new cases of prostate cancer and 27,540 deaths by PCa, making this disease the second leading cause of cancer-related death for North American men.

Men with PCa may develop lower urinary tract symptoms (LUTS) when prostate tumors invade or compress the prostatic urethra, the bladder or the neurovascular bundles, or when the prostate is enlarged. It has been estimated that over 40% of men with PCa experience moderate or severe LUTS. LUTS can impact profoundly on a man's quality of life (QoL); an effect that increases with increasing LUTS severity.

Transurethral resection of prostate (TURP) can offer immediate relief of the obstruction in patients with benign prostatic hyperplasia (BPH). In contrast, palliative TURP (p-TURP) (the so-called "channel" TURP), is transurethral resection of prostate tissue in a patient with metastatic or locally advanced and/or previously treated PCa to alleviate obstructive voiding symptoms.

Al¬though TURP is commonly performed to relieve bladder outlet ob¬struction (BOO) symptoms in patients with BPH, little known about the outcome of palliative transurethral plasma kinetic resection of prostate (p-TUPKRP) in patients with ad-vanced PCa.

Gonadotropin-releasing hormone (GnRH) agonists as androgen deprivation therapy (ADT) are the standard treatment for many patients with PCa, particularly those with advanced or metastatic disease. The impact of ADT on tumor control and achieving the reduction in prostate specific antigen (PSA) is well established. But there is less information available on the effects on LUTSs in men with PCa. Some short-term studies of ADT with the GnRH antagonist or with ADT in the neoadjuvant setting have demonstrated reductions in LUTSs, measured by the International Prostate Symptom Score (IPSS). There are few published data on the longer-term effects of ADT on LUTSs, apart from an earlier interim analysis of data from the current study.

In this study, p-TUPKRP combined with ADT will perform for 50 patients with advanced PCa complicated with severe LUTS. As a control, other 50 advanced PCa patients with same symptoms will be treated with ADT only. Some clinical data, including PSA, IPSS, QoL, Urinary flow rate (UFR), ECOG Score, Overall survival (OS), progression-free survival (PFS), will be analyzed. It is expected to explore the efficacy and safety of the combination therapy to advanced PCa with severe LUTS.

ELIGIBILITY:
Inclusion Criteria:

1. Hormone sensibility advanced prostate adenocarcinoma, clinical stages are T3-4N0-1M0-1b；
2. International prostate symptom score is equal to or greater than 20;
3. Maximum flow rate is equal to or less than 10ml/s, or bladder outlet obstruction is diagnosed by urodynamics
4. Any of the following complication: ① calculus in bladder; ② Recurrent urinary tract infections; ③Inguinal hernia; ④vesicoureteral reflux
5. The physical status score of the Eastern Cancer Cooperative Group (ECOG) is 0 or 1;
6. There has been no previous evidence of malignancy in the past five years.
7. The patient is in good physical condition and able to tolerate anesthesia and surgery;
8. There are no allergic reactions and liver or kidney function damage to endocrine drugs;
9. Ability to take and retain medicines;
10. Ability to follow study visit schedules and other program requirements；
11. Be able to understand the character and purpose of the study, including possible risks and side effects; Be able to work with researchers and follow the requirements of the entire study;
12. Ability to sign and date informed of the full character and purpose of the study, including possible risks and side effects, and sufficient time and opportunity to read and understand the information about this study.

Exclusion Criteria:

1. Patients with castration-resistant prostate cancer;
2. The physical status score of East Cancer cooperative Group is equal to or greater than 2;
3. There has been previous evidence of other malignancy in the past five years;
4. Patients with high coagulation and cannot stop taking anticoagulants;
5. Abnormal coagulation function such as hemophilia;
6. The patients are in poor physical condition and cannot tolerate anesthesia and surgery;
7. The patients have allergy or toxic side effects and other adverse reaction to endocrine drug;
8. Patients with active tuberculosis or other fulminating infectious disease;
9. Patients with immunodeficiency;
10. Patients with the lower limb and joint function abnormality, cannot maintain the lithotomy position for a long time;
11. Patients with urethral stricture;
12. Unable to comply with study visit schedule and other program requirements;
13. Any patients, who are regarded cannot not participate in the study;

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
PSA | 3 months
  Prostate specific antigen, or PSA, is a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA test measures the level of PSA in a man's blood. For this test, a blood sample is sent to a laboratory for analysis. The results are usually reported as nanograms of PSA per milliliter (ng/mL) of blood. The blood level of PSA is often elevated in men with prostate cancer. PSA will be used to evaluate the effectiveness of tumor therapy
Maximum flow rate | 3 months
  Uronary flow rate is the volumetric flow rate of urine during urination. It is a measure of the quantity of urine excreted in a specified period of time (per second or per minute). It is measured with uroflowmetry, a type of flowmetry. The "Q" (a conventional symbol for flow rate) is used as a symbol for urine flow rate. Qmax indicates the maximum flow rate. Qmax is used as an indicator for the diagnosis of enlarged prostate. A lower Qmax may indicate that the enlarged prostate puts pressure on the urethra,
IPSS | 3 months
  International prostate symptom score(IPSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35. The first seven questions of the I-PSS are identical to the questions appearing on the American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows: Mild (symptom score less than of equal to 7); Moderate (symptom score range 8-19); Severe (symptom score range 20-35).
QoL | 3 months
  Quality of life due to urinary symptoms is base on the question, If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? The International Scientific Committee (SCI), under the patronage of the World Health Organization (WHO) and the International Union Against Cancer (UICC), recommends the use of only a single question to assess the quality of life. The answers to this question range from "delighted" to "terrible" or 0 to 6. Although this single question may or may not capture the global impact of benign prostatic hyperplasia (BPH) Symptoms or quality of life, it may serve as a valuable starting point for a doctor-patient conversation.
ECOG | 3 months
  Physical status scores of East Cancer cooperative Group. Grade 0:Fully active, able to carry on all pre-disease performance without restriction; Grade 1:Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; Grade 2:Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; Grade 3:Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; Grade 5: dead.
MRI | 6 months
  Magnetic Resonance Imaging (MRI) of the prostate uses a powerful magnetic field, radio waves and a computer to produce detailed pictures of the structures within a man's prostate gland. It is primarily used to evaluate the extent of prostate cancer and determine whether it has spread. MRI of the prostate can be used to determine the efficacy of therapy and imaging progression-free survival.
SPECT | 6 months
  In prostate cancer, bone is the second most common site of metastatic disease after lymph nodes. Single-Photon Emission Computed Tomography (SPECT) in imaging bone metastases is increasing in popularity for staging newly diagnosed prostate cancer and for assessing response to therapy. SPECT can be used to determine the efficacy of therapy and imaging progression-free survival.
PVR | 3 months
  PVR is post void residual urine volume. In those who can void, incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal.
OS | 12 months
  Overall survival, or OS, the length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, that patients diagnosed with the disease are still alive.
PFS | 12 months
  Progression-free survival (PFS) is "the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse"

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Huang, MD, Study Director — The Third Xiangya Hospital of Central South University